CLINICAL TRIAL: NCT05689801
Title: Pilot Study: Describe the Effect of the Optimized Hemodialysis Technique (HDx) With Medium Cut-Off Membrane on Recovery Time and Quality of Life
Brief Title: Describe the Effect of the Optimized Hemodialysis Technique (HDx) With Medium Cut-Off Membrane on Recovery Time and Quality of Life
Acronym: EHDXTRQV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A01511-42
Record Dates: First submitted 2022-12-22; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Terminal Renal Insufficiency
Keywords: terminal renal insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient on conventional hemodialysis then on optimized hemodialysis (Experimental)
  Interventions: Other: Questionnaire "recovery time after a dialysis session".; Other: SF-12 questionnaire; Other: EQ-5D-5L Questionnaire; Other: Pittman, John et McIntyre questionnaire; Procedure: Conventional hemodialysis; Procedure: Optimized hemodialysis

INTERVENTIONS:
Other: Questionnaire "recovery time after a dialysis session". — A very short questionnaire just after the dialysis session
Other: SF-12 questionnaire — Questionnaire about quality of life of the patient
Other: EQ-5D-5L Questionnaire — Questionnaire about quality of life of the patient
Other: Pittman, John et McIntyre questionnaire — Questionnaire about quality of life of the patient under dialysis
Procedure: Conventional hemodialysis — patient on polyethersulfone membrane dialysis (Revaclear®, Baxter) with HemoControl™ for 12 weeks
Procedure: Optimized hemodialysis — patient on Medium Cut-Off membrane dialysis (Theranova®, Baxter) with HemoControl™ for 12 weeks.

SUMMARY:
In this study, the effect of optimizing the dialytic technique using simple questionnaires carried out in clinical routine will be described.

More specifically, the conventional dialysis technique will be combined with biofeedback software called HemoControl™. The recovery time and quality of life of patients who will use a polyethersulfone membrane (Revaclear®) and a Medium Cut-Off (MCO) membrane (Theranova®) will be observed.

The main objective is to describe the evolution of recovery time after a dialysis session in conventional hemodialysis (HD) on Revaclear® membrane and in so-called optimized hemodialysis (HDx) on MCO membrane, Theranova®.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female (using contraceptives, if of childbearing age), over 18 years of age
* Patient on conventional hemodialysis with synthetic membrane for at least 3 months
* Patient with a recovery time after the dialysis session ≥ 4 hours
* Informed patient who has signed a written consent to participate in the study
* Affiliated patient or beneficiary of a social security scheme

Exclusion Criteria:

* Patient whose seniority of dialysis is less than 3 months
* Pregnant woman
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Patient with severe cognitive impairment
* Medically unstable or frail patient
* Patient who did not sign an informed consent form accepting this research (refusal of consent or absence of signature).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-06-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Result of the questionnaire "recovery time after a dialysis session" | 7 months
  only one question : how long time recovering after a dialysis session (hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Claude Galien, Quincy-sous-Sénart, France